CLINICAL TRIAL: NCT05079412
Title: Does Non-Invasive Ventilation Neurally-Adjusted Ventilatory Assist (NIV-NAVA) Improve Diaphragmatic Function in Preterm Infants?
Brief Title: Does NIV-NAVA Improve Diaphragmatic Function in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Adel Mohamed, Principal Investigator, Mount Sinai Hospital, Canada
Other Study IDs: 19-0324-E
Record Dates: First submitted 2021-09-30; First posted 2021-10-15 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Disease
Keywords: preterm; neonates; Ultrasound; non-invasive; ventilation; Diaphragm; Lung; NIV-NAVA; NIPPV
MeSH Terms: conditions — Respiration Disorders; Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NIV-NAVA group: Premature infants (22 0/7 to 29 6/7 weeks gestation) with respiratory distress syndrome who are admitted to Mount Sinai NICU and are supported by NIV-NAVA for at least 24 hours are enrolled in this arm after obtaining parents' consent.
  Interventions: Other: Chest ultrasound
- NIPPV group: Premature infants (22 0/7 to 29 6/7 weeks gestation) with respiratory distress syndrome who are admitted to Mount Sinai NICU and are supported by NIPPV for at least 24 hours are enrolled in this arm after obtaining parents' consent.
  Interventions: Other: Chest ultrasound

INTERVENTIONS:
Other: Chest ultrasound — Chest ultrasound will be performed to eligiable (consented) patient after being on the respiratory support (NIV-NAVA vs NIPPV) for at least 24 hours. Both diaphragmatic function and lung ultrasound score will performed. Investigator interpreting the scans will be blind to patients type of respiratory support or clinical status.

SUMMARY:
Non-Invasive Positive Pressure Ventilation (NIPPV) provides un-synchronized positive pressure and considered to be superior to nCPAP in preventing extubation failure. Recently, Non-Invasive Ventilation Neurally-Adjusted Ventilatory Assist (NIV-NAVA) was introduced to NICU. NAVA is a ventilation mode that uses the electrical activity of the patient's diaphragm (Edi-signal) to guide both timing and magnitude of the support. However, it is unknown whether NIV-NAVA is superior to NIPPV in preventing extubation failure and preventing BPD.

Hence, the investigators aim to compare the effect of NIPPV and NIV-NAVA on diaphragm function in premature infants with RDS or evolving BPD. Our hypothesis is that infants treated with NIV-NAVA will have improved diaphragmatic function and lung scoring.

DETAILED DESCRIPTION:
STUDY POPULATION Premature infants with respiratory distress syndrome who are admitted to Mount Sinai NICU and are supported with NIPPV or NIV-NAVA.

Inclusion criteria

1. Infants that were born at 22 0/7 to 29 6/7 weeks gestation and admitted to the NICU at Mount Sinai Health System.
2. Infants that are on NIPPV or NIV-NAVA respiratory support for at least 24 hours at the time of enrolment.

Exclusion criteria

1. Infants with congenital anomalies.
2. Infants with known genetic disorder.
3. Infants with known lung malformation or diaphragm dysfunction.
4. Infants of whom parents declined consent.

Study Design and settings:

This is a prospective cohort study that includes premature infants born at 22 0/7 to 29 6/7 weeks GA in Mount Sinai Hospital and admitted to the NICU. Written consent will be obtained from parents or guardians prior to enrolment in the study. Enrolment of eligible infants will start after obtaining approval from Mount Sinai Research Ethics Board and parent's consent. Recruitment will be done over one year, and the investigators are expecting to recruit about 30 infants in the NIPPV group and similar number in the NIV-NAVA group.

Time of assessment; Eligible infants will be identified by a member of the infant's circle of care. Parents of infants who are eligible for the study will be approached for consent. Chest ultrasound (lung ultrasound and diaphragmatic function assessment) will be performed at > 7 days postnatally, provided that the infant is supported by either NIPPV or NIV-NAVA for at least 24 hours. CUS will be done prior to feeding to avoid any concerns of a full stomach on diaphragmatic assessment.

Study procedure: Functional assessment of the diaphragm combined with lung ultrasound examination will be done by one of the investigators.

Lung ultrasound assessment technique; Lung ultrasounds will be performed in a standardized manner. A longitudinal scan of the anterior and lateral chest walls will be performed. Three chest areas for each side (upper anterior, lower anterior, and lateral) will be assessed. Each area will have a score of 0 to 3 points with a total score between 0 to 18, which inversely correlates with lung aeration.

Diaphragmatic assessment technique; Diaphragm assessment will be performed in the supine position. To measure diaphragmatic excursion, the curvilinear probe will be placed on the lower intercostal spaces between the mid-clavicular and anterior axillary lines on the right side and between the anterior and mid-axillary lines for the left side. Using the B mode, the proper exploration line of the diaphragm will be detected by directing the beam perpendicular to the posterior third of the right hemidiaphragm. By M mode, the cyclic caudal diaphragmatic displacement with respiration will be measured as the perpendicular distance between the most caudal point of the liver or spleen at the end of expiration and the end of inspiration. The average of three respiratory cycles will be taken.

The assessment of the diaphragmatic efficiency as a pressure generator will be evaluated using the diaphragmatic thickness fraction. Diaphragmatic thickness will be measured at the apposition zone which can be obtained by placing the linear transducer above the 10th rib in the mid-axillary or anterior axillary lines in the right intercostal spaces. By B mode, three distinct layers will be seen, the diaphragm as a hypo-echoic area bordered by two clear echogenic lines of the pleural membrane (upper line) and the peritoneal membrane (lower line). Using M-mode tracing, inspiratory diaphragmatic thickness will be measured as the maximum perpendicular distance between pleural and peritoneal layers and by the same way expiratory diaphragmatic thickness will be recorded. diaphragmatic thickness fraction will be calculated using the following formula:

diaphragmatic thickness fraction = [(inspiratory thickness - expiratory thickness)/expiratory thickness] x 100.

The average of the calculated diaphragmatic thickness fraction from three respiratory cycles will be estimated. The higher scores the better the diaphragmatic function. All Chest ultrasound assessments will be undertaken using a standard aseptic technique.

ELIGIBILITY:
Inclusion criteria

1. Infants that were born at 22 0/7 to 29 6/7 weeks gestation and admitted to the NICU at Mount Sinai Health System.
2. Infants that are on NIPPV or NIV-NAVA respiratory support for at least 24 hours at the time of enrolment.

Exclusion Criteria:

1. Infants with congenital anomalies.
2. Infants with known genetic disorder.
3. Infants with known lung malformation or diaphragm dysfunction.
4. Infants of whom parents declined consent.

Ages: 2 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants that were born between 22 0/7 to 29 6/7 weeks gestation and were admitted to the NICU at Mount Sinai Health System will be eligible for the study. Infants will be enrolled after obtaining parents' consent and Research Ethics Board approval
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the diaphragmatic Thickness (in millimetre) in neonates on each arm (NIV-NAVA and NIPPV) | 1 YEAR
  Chest ultrasound will be performed to eligible (consented) patient after being on the respiratory support (NIV-NAVA vs NIPPV) for at least 24 hours. diaphragmatic Thickness (in millimetre) will be measured. Investigator interpreting the scans will be blind to patients type of respiratory support or clinical status.
Evaluation of the diaphragmatic excursion (in millimetre) in neonates on each arm (NIV-NAVA and NIPPV) | 1 YEAR
  Chest ultrasound will be performed to eligible (consented) patient after being on the respiratory support (NIV-NAVA vs NIPPV) for at least 24 hours. diaphragmatic Excursion (in millimetre) will be measured. Investigator interpreting the scans will be blind to patients type of respiratory support or clinical status.

SECONDARY OUTCOMES:
Lung ultrasound score for infants in NIV-NAVA group vs NIPPV group | 1 YEAR
  Chest ultrasound will be performed to eligible (consented) patient after being on the respiratory support (NIV-NAVA vs NIPPV) for at least 24 hours. Lung ultrasound score will performed. Lung ultrasound score range from 0 to 18 points. while 0 points (good score) means normal lung, 18 points (bad score) mean severely affected lung. Investigator interpreting the scans will be blind to patients type of respiratory support or clinical status.

CONTACTS AND LOCATIONS:
Overall Officials: Adel Mohamed, MD, Principal Investigator — Mount Sinai Hospital- Toronto, ON, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Elkhouli M, Tamir-Hostovsky L, Ibrahim J, Nasef N, Mohamed A. Ultrasonographic assessment of diaphragmatic function in preterm infants on non-invasive neurally adjusted ventilatory assist (NIV-NAVA) compared to nasal intermittent positive-pressure ventilation (NIPPV): a prospective observational study. Eur J Pediatr. 2023 Feb;182(2):731-739. doi: 10.1007/s00431-022-04738-8. Epub 2022 Dec 2. PMID 36459227